CLINICAL TRIAL: NCT04450433
Title: Functional Study of Metabolites in Patients With Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Liuhuadong's Research Group
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Baseline table of patients
  Interventions: Diagnostic Test: aortic dissection and healthy people
- Differential metabolites of two groups of control patients
  Interventions: Diagnostic Test: aortic dissection and healthy people
- Functional verification of differential metabolites
  Interventions: Diagnostic Test: aortic dissection and healthy people

INTERVENTIONS:
Diagnostic Test: aortic dissection and healthy people — Differential expression of metabolites in patients with aortic dissection and healthy people

SUMMARY:
Research on metabolites in patients with aortic dissection, with a view to finding products with high or low metabolism in patients with aortic dissection, looking for metabolic factors related to the onset of aortic dissection, and further verifying the role of metabolic factors in disease through functional verification The role of formation, and ultimately explore the early screening of potential aortic dissection patients

ELIGIBILITY:
Inclusion Criteria:

* patients with Aortic dissection

Exclusion Criteria:

* Sepsis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with aortic dissection and 15 healthy people
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Differential expression of metabolites in two groups of patients | 2019-11----2021.01
  Differential expression of metabolites in the two groups of patients, looking for metabolic factors related to the incidence of aortic dissection, and further verifying the function of metabolites through functional methods, with a view to finding high-risk metabolic factors for patients with aortic dissection

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided